CLINICAL TRIAL: NCT07281950
Title: Dry Eye Surveys to Evaluate Acoltremon in Real World Treatment (DESERT)
Brief Title: Investigator Initiated Trial Using Dry Eye Surveys to Evaluate and Better Understand FDA Approved Acoltremon Treatment for Dry Eye Disease in Real World Treatment Settings (DESERT)
Acronym: (DESERT)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Center for Sight Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFS-DESERT-102
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye Disease (DED)
Keywords: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective, single-site, multi-location, single arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- all subjects meeing inclusion/exclusion will be dispensed FDA Approved acoltremon (Other): all subjects meeing inclusion/exclusion will be dispensed FDA Approved acoltremon 0.003%
  Interventions: Drug: acoltremon 0.003%

INTERVENTIONS:
Drug: acoltremon 0.003% — single arm

SUMMARY:
Dry eye disease (DED) is a common, chronic and multifactorial disease of the ocular surface presenting with signs and symptoms of ocular discomfort, visual disturbance and fluctuation, tear film instability, ocular surface inflammation and damage.

It significantly affects patients' quality of life and is one of the most frequent reasons for visits to eye care providers. Many patients remain symptomatic in real-world settings despite current pharmacologic therapeutic options available. As symptoms often lag behind ocular signs, a 3 month study with multiple time points has been designed to assess short term and mid-term symptomatic changes.

This study will use Dry Eye Surveys to evaluate Acoltremon in Real World Settings to help understand its real world effectiveness and potential to improve symptoms in dry eye patients.

DETAILED DESCRIPTION:
TRYPTYR (Acoltremon 0.003%) is a newly FDA approved therapy for dry eye disease with a novel mechanism of action. It is a TRPM8 receptor agonist that stimulates trigeminal nerve signaling, which has been associated with increased basal tear production. As randomized clinical trials are conducted under highly controlled conditions, their results may not fully represent the effectiveness of drugs in real-world settings.

Given TRYPTYR's (Acoltremon 0.003%) recent approval, there is a need to better understand how the medication performs in real-world settings and generate real-world evidence to assess its effectiveness and impact on patient-reported symptoms in individuals with dry eye disease (DED). Real-world data is essential to evaluate treatment outcomes in routine clinical practice. The SPEED (Standard Patient Evaluation of Eye Dryness) questionnaire is a widely accepted clinical tool that captures the frequency and severity of DED symptoms from the patient's perspective. Incorporating the SPEED questionnaire into this study will enable a robust assessment of symptom burden and treatment-related changes, thereby addressing a critical unmet need in understanding TRYPTYR's real-world effectiveness and its potential to improve symptoms in DED patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults age 18 and older at Visit 1
* Have a previous history of dry eye disease, clinician diagnosed or self-reported, for at least 3 months
* Total SPEED score ≥ 6 on SPEED questionnaire at Visit 1 Screening & Baseline

Exclusion Criteria:

* History of ocular surgery (excluding LASIK or PRK) in the past 3 months
* History of LASIK or PRK in the past 12 months
* Initiation, discontinuation or change in dose of a systemic medication known to cause ocular drying (e.g., antihistamines or tricyclic antidepressants) less than 14 days prior to Visit 1 or a change in dosage is anticipated during the study.

  o Note: occasional short-term use of medications such as systemic antihistamines will be permitted provided that use was not within 24 hours of Visit 1 or anticipated use within 24 hours of any study visit.
* Active ocular infection or inflammation unrelated to dry eye disease (e.g., uveitis, blepharitis requiring antibiotics).
* Use of Restasis, Xiidra, Miebo, or any other topical anti-inflammatory medications within 30 days of Visit 1 and for the duration of the study.
* Use of varenicline nasal spray within 30 days of Visit 1 and for the duration of the study.
* Eyelid hygiene (such as "lid scrubs") is allowed but should be continued without change to current regiment at Visit 1 Baseline for the duration of the study.
* Use of other DED medications within 30 days of Visit 1 Baseline Use of artificial tears is allowed but must be preservative free and the dosing should not change from current regiment at Visit 1 Baseline.
* Use of amniotic membranes or serum tears within 90 days of Visit 1 Baseline
* Use of lid heating therapy (i.e., LipiFlow, iLUX, TearCare) within 90 days of Visit 1 Baseline and for the duration of the study.
* Punctal or intracanalicular plug inserted in either eyelid within 90 days prior to Visit 1 Baseline or anticipated plug insertion or occlusion at any time during the study.
* Current evidence of other significant ophthalmic disease requiring topical medication (e.g., glaucoma, ocular hypertension) or other disease the investigator believes may interfere with study findings or interpretation.
* Use of any topical ocular glaucoma medication within 30 days prior to the Screening visit or anticipated use during the study.
* Use of systemic medications that affect tear production (e.g., isotretinoin, antihistamines) unless on stable doses for > 30 days.
* Severe ocular surface disease or damage (e.g., corneal ulcers, neurotrophic keratopathy).
* Have had a corneal transplant in either or both eyes.
* Use of contact lenses in either eye within 7 days prior to the Baseline visit or planned use during the study and unwilling to discontinue use during the duration of the study.
* Known allergy or hypersensitivity to acoltremon or formulation ingredients.
* Current pregnancy or breastfeeding
* Women of childbearing potential who are not using an acceptable means of contraception. Acceptable means of contraception include hormonal contraceptives (i.e. oral, implantable, injectable, or transdermal contraceptives, with a barrier such as a diaphragm or a condom) or intrauterine devices. For non-sexually active females, abstinence may be regarded as an adequate method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
• Mean Change in SPEED questionnaire score at 1 month (day 30 ± 3 days) | Mean Change in SPEED questionnaire score at 1 month (day 30 ± 3 days)
  Mean Change in SPEED questionnaire score at 1 month (day 30 ± 3 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sight, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not plan to share individual participant data due to concerns about participant privacy and confidentiality.